CLINICAL TRIAL: NCT00538421
Title: Opioid-potentiated Volative Anaesthetic(Sevoflurane)Compared to Remifentanil and Propofol During Abdominal Aortic Aneurysm Surgery
Brief Title: Opioid-potentiated Volative Anaesthetic Vs. Remifentanil And Propofol During Abdominal Aortic Aneurysm Surgery
Acronym: ABSENT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sykehuset i Vestfold HF (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Espen Lindholm, Chief consultant, Sykehuset i Vestfold HF
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-07294b (REK); 2007-000002-79 (Eudract); 17089 (NSD)
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Aortic Diseases; Abdominal; Aneurysm; Surgery
Keywords: propofol; Anaesthesia; Sevoflurane; Abdominal; Aortic; Aneurysm
MeSH Terms: conditions — Aortic Diseases; Aneurysm | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Propofol
- 2 (Active Comparator)
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Infusion intravenously (IV) 0-10 mg/kg/h
  Arms: 1
Drug: Sevoflurane — 0,7-1,5 MAC
  Arms: 2

SUMMARY:
Comparing 2 different anaesthetic methods during abdominal aortic aneurysm surgery. The patients will be followed up 30 days postoperative. Number of patients included will be 200. Perioperative details will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for open, elective abdominal aortic aneurysm surgery.
* ASA group 1-4.

Exclusion Criteria:

* Patients below 18 years.
* Patients who are included in other pharmaceutical studies.
* Opioids-, benzodiazepins-, antiepileptic drugs-, alcohol- and α2-agonists abuse.
* Pregnant and breastfeeding women.
* Patients with familiar history of malignant hyperthermia.
* Patients with known hypersensitivity for opioids, propofol or volative anaesthetics.
* Patients with considerable arrythmia (atrial fibrillation /atrial flutter is acceptable). Uncontrolled hypertension, serious psychiatric disease.
* Patients with unstable angina pectoris or myocardial infarction last month before inclusion.
* Acute abdominal aortic surgery. Acute dissection or rupture.
* Planned laparoscopic abdominal aortic aneurysm surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2008-03; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Espen Lindholm, MD, Study Director — Sykehuset i Vestfold HF
Locations (1):
- Sykehuset i Vestfold HF, Tønsberg, Norway